CLINICAL TRIAL: NCT06605261
Title: Effect of Yoga Program on Quality of Life in Women With Breast Cancer Receiving Endocrine Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gözde Gür (Other)
Responsible Party: Sponsor-Investigator, Gözde Gür, Lecturer, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-10/453
Record Dates: First submitted 2024-09-16; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Yoga; Quality of Life; Nursing; Endocrine Therapy
Keywords: breast cancer; yoga; quality of life; nursing; endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Yoga; Methods; Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (intervention) Group (Experimental): A yoga program will be conducted with 64 women undergoing endocrine therapy, experiencing joint pain or vasomotor symptoms, who are randomly assigned to the intervention group. The program will be delivered online via a digital platform for 4 weeks, 60 minutes per session, 4 days a week, with an instructor. An introductory session will provide information on yoga philosophy and program details. Each session will start with breathing exercises (pranayama), followed by yoga postures (asanas), and end with meditation. Participants will receive a yoga guide and necessary equipment (yoga mats, blocks) before starting. The FACT-ES Endocrine Symptoms Subscale will be re-administered in the second week. After each session, participants will report any adverse effects via digital communication. One month after the program, participants will be asked if they continued yoga at home, and reasons for discontinuation will be recorded.
  Interventions: Other: Yoga (intervention) group
- Control Group (No Intervention): No intervention will be applied to individuals in this group, and they will continue with the routine exercises recommended by their physicians. After their data is collected as part of the control group, they will be invited by the researcher to participate in the online yoga sessions conducted with the intervention group.

INTERVENTIONS:
Other: Yoga (intervention) group — The yoga (intervention) group comprises 64 women with breast cancer who have been randomly assigned and are undergoing endocrine therapy. To alleviate arthralgia and vasomotor symptoms (hot flashes, night sweats), a structured yoga program will be administered during the initial months of endocrine therapy, consisting of 60-minute sessions, 4 days per week, for a duration of one month.
  Arms: Yoga (intervention) Group

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effect of a yoga program on improving the quality of life, reducing joint pain, and alleviating vasomotor symptoms (night sweats, hot flashes) in women with breast cancer undergoing endocrine therapy.

The main questions it aims to answer are:

Does the yoga program significantly improve the quality of life in women with breast cancer undergoing endocrine therapy? Is the yoga program effective in reducing joint pain in women with breast cancer? Does the yoga program reduce the severity of night sweats and hot flashes in women with breast cancer? Researchers will compare the intervention group, which will receive the yoga program, to the control group, which will continue with their physician-recommended routine exercise, to see if there is a difference in these outcomes.

Participants will: Participants will consist of women with breast cancer undergoing endocrine therapy, with 64 in the yoga (intervention) group and 64 in the control group.

Complete the;Patient Assessment Form; and the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) scale.

The intervention group will participate in a 60-minute yoga program, delivered online via a digital platform, four days a week for four weeks, led by an instructor.

The control group will not receive any intervention and will continue with their physician-recommended routine exercise.

DETAILED DESCRIPTION:
The goal of this randomized controlled trial is to evaluate the effect of a yoga program on improving the quality of life, reducing joint pain, and alleviating vasomotor symptoms (such as night sweats and hot flashes) in women with breast cancer undergoing endocrine therapy. The participants will be divided into two groups: 64 women in the yoga (intervention) group and 64 women in the control group.

Hypotheses:

H1: The yoga program will significantly improve the quality of life in women with breast cancer undergoing endocrine therapy.

H1: The yoga program will be effective in reducing joint pain in women with breast cancer.

H1: The yoga program will be effective in reducing the severity of night sweats and hot flashes in women with breast cancer.

Population:

The study population consists of women who have completed surgical treatment in oncology units, have completed chemotherapy or radiation therapy, and have recently started adjuvant endocrine therapy. The sample size, calculated using G power with an effect size of 0.5, a 5% error margin, and 80% power, includes 128 participants (64 in the intervention group and 64 in the control group), taking into account possible data losses.

Data Collection Tools:

The research data will be collected using the; Patient Identification Form and the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) scale.

Patient Identification Form: Developed by the researcher based on literature, this form consists of two sections. The first section includes personal characteristics such as age, gender, education level, and body mass index. The second section investigates medical history, general health information, and lifestyle habits (e.g., smoking, alcohol use, diet, and sleep patterns).

Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES): This comprehensive scale was developed to evaluate the quality of life of cancer patients, particularly those receiving endocrine therapy. The scale consists of 46 items rated on a scale from 0 to 4, and it includes five main subscales: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Endocrine Symptom Subscale. Some negatively worded items are reverse-scored, and raw scores are totaled. Subscale scores are calculated separately, and the total score is the sum of the subscale scores. Higher scores indicate better quality of life and fewer symptoms. The scale can be scored manually, and appropriate prorating methods are applied in the case of missing data. It is valid for cancer patients aged 18 and over, assessing experiences over the past seven days. The assessment is conducted using a 5-point Likert scale and takes approximately 10-15 minutes. It can be administered both in paper form and electronically, and completed via self-reporting or interviews if necessary.

Process:

Participants in both the intervention and control groups will be informed about the purpose and steps of the study, and the Informed Consent Form will be read and signed. Written and verbal consent will be obtained from those who agree to participate in the study. In the initial phase, data will be collected via face-to-face interviews using the Patient Assessment Form along with weight measurement and basic movements (e.g., standing while touching toes for 30 seconds, raising arms overhead, moving from standing to sitting position). The FACT-ES scale will also be administered during this interview. Data collection will continue using digital communication tools every two weeks once the online yoga program begins.The intervention group will participate in a 60-minute yoga program, delivered online via a digital platform, four days a week for four weeks, led by an instructor. The control group will not receive any intervention and will continue with their physician-recommended routine exercise.

Yoga Program (Intervention Group):

Participants in the intervention group will participate in a 60-minute yoga program, delivered online via a digital platform, four days a week for four weeks.

Each session will begin with breathing exercises (pranayama), followed by yoga postures (asanas), and end with meditation.

While the yoga program continues, the Endocrine Symptoms Subscale of the FACT-ES scale will be applied in the 2nd week.

Since the program is conducted online, participants will be advised to perform yoga in a quiet and hygienic environment conducive to practice.

Before starting the yoga practice, participants will be provided with a yoga guide by the researcher.

An introductory session will be held to explain the philosophy of yoga and the details of the program.

Yoga mats, blocks, and other necessary equipment will be provided to participants before starting the practice.

After each yoga session, participants will be asked to provide feedback on any adverse effects they may have experienced, which will be recorded through digital communication tools.

One month after completing the four-week online yoga program, participants will be asked how often they have continued the yoga practice at home, and this will be recorded.

Participants who do not continue yoga practice will be asked to provide reasons, which will also be recorded.

Yoga Program Structure:

Warm-up (10 minutes) Pranayama (Breathing Exercise) - 5 minutes Dirga Pranayama (Three-Part Breath): Slows breathing and calms the mind. Gentle Neck Stretches - 5 minutes Relieves tension in the neck, where stress is often stored. Main Practice (45 minutes) Tadasana (Mountain Pose) - 5 minutes An excellent starting pose for improving posture and body awareness. Vrikshasana (Tree Pose) - 5 minutes Enhances balance and focus, strengthens the legs. Baddha Konasana (Butterfly Pose) - 5 minutes Increases flexibility in the hips and inner thighs, relieves the pelvic area. Marjaryasana-Bitilasana (Cat-Cow Stretch) - 5 minutes Stretches and revitalizes the spine, alleviates back pain. Paschimottanasana (Seated Forward Bend) - 5 minutes Stretches the back and legs, reduces stress and fatigue. Bhujangasana (Cobra Pose) - 5 minutes This chest-opening pose increases respiratory capacity and strengthens the spine.

Balasana (Child Pose) - 5 minutes Provides deep relaxation and stress reduction. Supta Matsyendrasana (Reclined Twist) - 5 minutes Stretches and relaxes the spine, soothes the digestive system. Cool-Down (10 minutes) Supta Baddha Konasana (Reclined Butterfly Pose) - 5 minutes

* Provides deep relaxation and gently stretches the inner thighs. Savasana (Corpse Pose) - 5 minutes
* Promotes deep relaxation and mental clarity.

Data Analysis: The data obtained from the study will be analyzed using the IBM SPSS Statistics 23 (IBM SPSS, Turkey) software. To test for the normality of the data distribution, the Kolmogorov-Smirnov test will be used. Values with skewness and kurtosis between ±2.0 will be considered to have a normal distribution. Descriptive statistics such as mean, standard deviation, percentage, and frequency will be used. If the data show a parametric distribution, One-Way Analysis of Variance (ANOVA) will be used for comparisons between more than two groups, and Repeated Measures ANOVA will be applied for repeated measurements. To determine the differences in quality of life scores between groups, an independent samples t-test will be conducted. If the data do not show a normal distribution, the Mann-Whitney U test will be applied. In addition, the Chi-Square test will be used to evaluate sociodemographic differences. A significance level of p will be considered the threshold for statistical significance. Finally, Cohen d will be calculated to evaluate effect size.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Having the ability to read, write, and speak Turkish,
* Having a diagnosis of breast cancer,
* Having completed surgical treatment,
* Having completed chemotherapy or radiation therapy,
* Recently starting endocrine therapy,
* Having a Body Mass Index (BMI) below 35.

Exclusion Criteria:

* Being over 70 years of age,
* Having a diagnosis of metastatic disease,
* Previous participation in yoga or similar exercises,
* Having a physical disability that prevents practicing yoga,
* Having a condition that causes shortness of breath (e.g., COPD),
* Having another chronic heart or lung disease that prevents yoga practice,
* Having a serious psychiatric illness or cognitive impairment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) | 1 week before the participants start the Yoga program.
  Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES): This comprehensive scale was developed to evaluate the quality of life of cancer patients, particularly those receiving endocrine therapy. The scale consists of 46 items rated on a scale from 0 to 4, and it includes five primary subscales: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Endocrine Symptom Subscale. Subscale scores are calculated separately, and the total score is the sum of the subscale scores. Higher scores indicate better quality of life and fewer symptoms. It is valid for cancer patients aged 18 and over, assessing experiences over the past seven days. The assessment uses a 5-point Likert scale and takes approximately 10-15 minutes.
Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) | through study completion, average of one year
  Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES): This comprehensive scale was developed to evaluate the quality of life of cancer patients, particularly those receiving endocrine therapy. The scale consists of 46 items rated on a scale from 0 to 4, and it includes five primary subscales: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Endocrine Symptom Subscale. Subscale scores are calculated separately, and the total score is the sum of the subscale scores. Higher scores indicate better quality of life and fewer symptoms. It is valid for cancer patients aged 18 and over, assessing experiences over the past seven days. The assessment uses a 5-point Likert scale and takes approximately 10-15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Gür, MSc, Principal Investigator — İstanbul University Cerrahpaşa; Aysun Ardıç, Assoc Prof, Principal Investigator — İstanbul University Cerrahpaşa

IPD SHARING:
Plan to Share IPD: No